CLINICAL TRIAL: NCT06248866
Title: Effect Of Extracorporeal Shock Wave Therapy On Ultrasonography Changes In Patients With Palmar Fibromatosis: A Randomized Controlled Trial
Acronym: ESWT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nabil Mahmoud Ismail Abdel-Aal, principle investigator nabil mahmoud ismail abdel-aal, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004965
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Palmar Fibromatosis
Keywords: Extracorporeal Shock Wave Therapy; Ultrasonography Changes; Palmar Fibromatosis
MeSH Terms: conditions — Dupuytren Contracture | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: extracorporeal shock wave therapy and traditional treatment
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extracorporeal Shock Wave Therapy (Experimental): patients will receive Extracorporeal Shock Wave Therapy and traditional treatment three times a week for six weeks
  Interventions: Other: Extracorporeal Shock Wave Therapy; Other: traditional treatment
- traditional treatment (Active Comparator): patients will receive traditional treatment three times a week for six weeks
  Interventions: Other: traditional treatment

INTERVENTIONS:
Other: Extracorporeal Shock Wave Therapy — The affected hand or fingers will be positioned comfortably to ensure optimal access to the fibromatosis lesion. Gel or oil will be applied to the skin to enhance the transmission of shock waves. Shock wave therapy will be administered using the selected energy level and frequency settings. Energy level and frequency will be customized based on individual patient requirements. (1000-1500 shock/session, frequency between 5-12HZ, compression power of 1.5- 2.5 bars).and will receive traditional treatment
  Arms: Extracorporeal Shock Wave Therapy
Other: traditional treatment — the patients will receive traditional treatment in the form of laser (A low-level laser device with a wavelength of 830 nm and power output of 50 mW will be used as one Of the pain relief methods), ultrasound (An ultrasound device with a frequency of 1 MHz and an intensity of 1.5 W/cm² will be used), stretching and strengthening exercise and splinting.

SUMMARY:
this study will be conducted to investigate the effect of extracorporeal shock wave therapy on ultrasonography chnges In patients with palmar fibromatosis

DETAILED DESCRIPTION:
Palmar fibromatosis, also known as Dupuytren's contracture, is a condition that affects the hand and fingers. It is characterized by the thickening and tightening of the fascia, a layer of connective tissue beneath the skin of the palm. This thickening and tightening can lead to the formation of nodules or cords that restrict the movement of the affected fingers. The treatment options for palmar fibromatosis vary depending on the severity of the condition and its impact on hand function. Mild cases may not require immediate treatment but should be regularly monitored. However, if the symptoms worsen or hinder hand function, there are several treatment options available. Extracorporeal shock wave therapy (ESWT) is a non-invasive physical therapy procedure that uses high-energy sound waves to treat various musculoskeletal conditions. It is commonly used to manage pain and promote healing in conditions such as plantar fasciitis, tendinitis, calcific tendinitis, and other similar disorders The ESWT has shown promising results in reducing pain, improving function, and promoting healing in various musculoskeletal conditions. sixty patients with palmar fibromatosis will be assigned randomly to two groups; first one will receive extracorporeal shock wave with traditional therapy and the other one will receive traditional therapy only

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with palmar fibromatosis.
* Adults aged 18 to 70 years.
* Patients of any stage of physiological change of the disease (nodules cords and contractures).

Exclusion Criteria:

* Patients with contraindications to extracorporeal shock wave therapy.
* Patients with a history of previous surgery for palmar fibromatosis.
* Patients with comorbidities or conditions that may affect the outcomes of the study.
* Patients of ganglions and palmar tendon fibrosis.
* Patients of sever and morbid obesity.
* End stage disease with psychological disturbance nature.
* Pregnant women.
* Cardiac and pulmonary unstable patients may affect results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-10 (Estimated); Primary Completion 2024-07-10 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
thickness of lesion | up to six weeks
  Ultrasonography will be used to assess the thickness of lesion

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder, and Hand | up to six weeks
  The Arabic version of the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire will be administered to evaluate functional outcomes.The questionnaire consists of 11 items related to daily activities and symptoms. Each item is rated on a 5-point Likert scale, with higher scores indicating greater disability
pressure pain threshold | up to six weeks
  algometer will be used to assess pressure pain threshold
hand grip strength | up to six weeks
  Jamar hand held dynamometer will be used to assess hand grip strength
finger range of motion | up to six weeks
  goniometer will be used to assess finger range of motion